CLINICAL TRIAL: NCT06804850
Title: Neoadjuvant Low-Dose Radiotherapy Plus Targeted Therapy and Immunotherapy vs. Targeted Therapy Plus Immunotherapy in Resectable Head and Neck Squamous Cell Carcinoma: A Prospective Randomized Controlled Trial
Brief Title: Neoadjuvant Radiotherapy Plus Targeted Therapy and Immunotherapy vs. Targeted Therapy Plus Immunotherapy in Resectable HNSCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn prior to participant enrollment due to administrative and protocol optimization considerations.
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-196
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — tislelizumab; Immunotherapy; Afatinib; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Cohort (Experimental): 1. Tislelizumab administration on days 1 and 22, and afatinib continuous administration from days 1 to 42
  2. Low-dose radiotherapy, 4Gy/2f,radiotherapy using intensity-modulated radiotherapy technology.
  3. Standard of care surgery
  Interventions: Drug: Tislelizumab; Drug: Afatinib; Radiation: Low dose radiotherapy
- Control Cohort (Active Comparator): 1. Tislelizumab administration on days 1 and 22, and afatinib continuous administration from days 1 to 42
  2. Standard of care surgery
  Interventions: Drug: Tislelizumab; Drug: Afatinib

INTERVENTIONS:
Drug: Tislelizumab — 200mg IV Q3W
  Other Names: Immunotherapy
Drug: Afatinib — 30mg PO QD
  Other Names: Targeted therapy
Radiation: Low dose radiotherapy — 4Gy / 2f. Intensity-modulated radiotherapy was used for radiotherapy.
  Other Names: Radiotherapy
  Arms: Treatment Cohort

SUMMARY:
This study compares the efficacy of neoadjuvant low-dose radiotherapy plus targeted-immunotherapy versus targeted-immunotherapy alone in resectable HNSCC patients.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is a common malignant tumor in the head and neck region. It has a high global incidence. Due to its special anatomical location, HNSCC affects patients' appearance and physiological functions. Comprehensive treatments such as surgery, radiotherapy, and chemotherapy are often adopted. More than 60% of patients are diagnosed with locally advanced or metastatic diseases, resulting in a low 5-year survival rate. Locally advanced patients have high recurrence and metastasis rates, and a poor prognosis. Neoadjuvant therapy before surgery theoretically can improve the possibility of radical surgery and the organ preservation rate. However, except for nasopharyngeal carcinoma, induction chemotherapy has not brought significant survival benefits to HNSCC patients, and new treatment regimens are urgently needed.

EGFR is overexpressed in 90% of HNSCC patients. The PD-1/PD-L1 signaling pathway is an important mechanism of tumor escape. Anti-PD-1/PD-L1 monoclonal antibodies have shown good efficacy and high safety in the treatment of malignant tumors. The combination of radiotherapy and immunotherapy can induce an anti-tumor immune response. Low-dose radiotherapy (LDRT) has low toxicity and can reprogram the tumor immune microenvironment. Multiple studies have confirmed the safety and feasibility of its combination with immunotherapy.

The previously conducted "Prospective, Single-arm Clinical Study of Low-dose Radiotherapy Plus Tislelizumab Combined with Afatinib for Neoadjuvant Therapy of Resectable Head and Neck Squamous Cell Carcinoma" has demonstrated good safety. Based on this, a head-to-head clinical study is planned to compare the efficacy of low-dose radiotherapy combined with targeted immunotherapy and pure targeted immunotherapy in patients with resectable head and neck squamous cell carcinoma, explore the clinical benefits of this new treatment measure, and provide new treatment options for HNSCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above.
2. Patients with pathologically confirmed HNSCC (except for nasopharyngeal carcinoma) and meet the following condition:

   ◦ were newly diagnosed and without distant metastasis; were deemed surgically
   * resectable evaluated by a head and neck surgeon;
   * were willing to undergo surgery.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Adequate organ and bone marrow function:

   * absolute neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 80 g/L, platelets ≥ 80 × 10^9/L;
   * ALT, AST and ALP < 2.5× upper limit of normal (ULN), total bilirubin ≤ 2×ULN; albumin≥ 2.8 g/dL；
   * creatinine clearance ≥ 60 ml/min；
   * INR≤ 1.5, APTT≤ 1.5×ULN.
5. Written informed consent.

Exclusion Criteria:

1. History of other malignancies (except for the history of malignant tumors that have been cured and have not recurred within 5 years, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, in situ cervical cancer, and gastrointestinal mucosal cancer, etc.）
2. Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
3. Any history of allergic disease, or a sever hypersensitivity reaction to drugs, or allergy to the study drug components.
4. Any of prior therapy with:

（1）anti-PD-1, anti-PD-L1/2, anti-CTLA-4 antibody, anti-EGFR antibody or EGFR-TKIs； （2）antitumor vaccine; （3）any active vaccine against an infectious disease within 4 weeks prior to the first dose or planned during the study period; （4）major surgery or serious trauma within 4 weeks before the first dose; toxicity from prior antitumor therapy has not recovered to ≤ CTCAE Version 5.0 Grade 1 or the level specified by the inclusion/exclusion criteria.

5. With serious medical diseases, such as grade II and above cardiac dysfunction (NYHA criteria), ischemic heart disease, supraventricular or ventricular arrhythmia, poorly controlled diabetes mellitus, poorly controlled hypertension, echocardiographic ejection fraction < 50%, etc.

6. With interstitial pneumonitis, non-infectious pneumonitis, active pulmonary tuberculosis, or history of pulmonary tuberculosis infection that were not controlled by treatment.

7. With hyperthyroidism, or organic thyroid disease. 8. With active infection, or unexplained fever during the screening period or 48 hours before the first dose.

9. With active hepatitis B or C, or known history of positive HIV test, or acquired immunodeficiency syndrome.

10. History of a clear neurological or psychiatric disorder. 11. History of drug abuse or alcohol abuse. 12. Women who are pregnant or breastfeeding, or have a reproductive plan from the screening period to 3 months after the end of the study, or have sex without contraceptive measures, or are unwilling to take appropriate contraceptive measures.

13. Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.

14. Any other factors that are not suitable for inclusion in this study judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response | Intraoperative
  Major Pathologic Response (MPR) was defined as fewer than 10% viable tumor cells.

SECONDARY OUTCOMES:
Pathologic Complete Response | Intraoperative
  Pathologic Complete Response (pCR) was defined as the absence of viable tumor cells.
Objective Response Rate | Up to 8 weeks
  Objective Response Rate (ORR) was defined as the percentage of participants with a best overall response of CR or PR using RECIST Criteria
Disease-free Survival | 1 year
  Disease-free Survival (DFS) was defined as the time from the administration of the first dose to first disease progression or death.
Progression-Free Survival | 1 year
  Progression-Free Survival (PFS) was defined as the time from the commencement of therapy to the first evidence of disease progression or death.
Overall Survival | 1 year
  Overall Survival (OS) was defined as the time from the start of treatment initiation to the patient's death from any cause.
Immune microenvironment | Intraoperative
  The local microenvironment of tumor cells, including the changes of T lymphocytes, B lymphocytes and other cells.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Pulte D, Brenner H. Changes in survival in head and neck cancers in the late 20th and early 21st century: a period analysis. Oncologist. 2010;15(9):994-1001. doi: 10.1634/theoncologist.2009-0289. Epub 2010 Aug 26. PMID 20798198
- [Background] Denaro N, Merlano MC, Russi EG. Follow-up in Head and Neck Cancer: Do More Does It Mean Do Better? A Systematic Review and Our Proposal Based on Our Experience. Clin Exp Otorhinolaryngol. 2016 Dec;9(4):287-297. doi: 10.21053/ceo.2015.00976. Epub 2016 Jun 25. PMID 27337948
- [Background] Harari PM. Promising new advances in head and neck radiotherapy. Ann Oncol. 2005;16 Suppl 6:vi13-vi19. doi: 10.1093/annonc/mdi453. PMID 15987991
- [Background] Haddad R, O'Neill A, Rabinowits G, Tishler R, Khuri F, Adkins D, Clark J, Sarlis N, Lorch J, Beitler JJ, Limaye S, Riley S, Posner M. Induction chemotherapy followed by concurrent chemoradiotherapy (sequential chemoradiotherapy) versus concurrent chemoradiotherapy alone in locally advanced head and neck cancer (PARADIGM): a randomised phase 3 trial. Lancet Oncol. 2013 Mar;14(3):257-64. doi: 10.1016/S1470-2045(13)70011-1. Epub 2013 Feb 13. PMID 23414589
- [Background] Cohen EE, Karrison TG, Kocherginsky M, Mueller J, Egan R, Huang CH, Brockstein BE, Agulnik MB, Mittal BB, Yunus F, Samant S, Raez LE, Mehra R, Kumar P, Ondrey F, Marchand P, Braegas B, Seiwert TY, Villaflor VM, Haraf DJ, Vokes EE. Phase III randomized trial of induction chemotherapy in patients with N2 or N3 locally advanced head and neck cancer. J Clin Oncol. 2014 Sep 1;32(25):2735-43. doi: 10.1200/JCO.2013.54.6309. Epub 2014 Jul 21. PMID 25049329
- [Background] Geoffrois L, Martin L, De Raucourt D, Sun XS, Tao Y, Maingon P, Buffet J, Pointreau Y, Sire C, Tuchais C, Babin E, Coutte A, Rolland F, Kaminsky MC, Alfonsi M, Lapeyre M, Saliou M, Lafond C, Jadaud E, Gery B, Zawadi A, Tourani JM, Khoury C, Henry AR, Hasbini A, Guichard F, Borel C, Meert N, Guillet P, Calais MH, Garaud P, Bourhis J. Induction Chemotherapy Followed by Cetuximab Radiotherapy Is Not Superior to Concurrent Chemoradiotherapy for Head and Neck Carcinomas: Results of the GORTEC 2007-02 Phase III Randomized Trial. J Clin Oncol. 2018 Nov 1;36(31):3077-3083. doi: 10.1200/JCO.2017.76.2591. Epub 2018 Jul 17. PMID 30016178
- [Background] Machiels JP, Haddad RI, Fayette J, Licitra LF, Tahara M, Vermorken JB, Clement PM, Gauler T, Cupissol D, Grau JJ, Guigay J, Caponigro F, de Castro G Jr, de Souza Viana L, Keilholz U, Del Campo JM, Cong XJ, Ehrnrooth E, Cohen EE; LUX-H&N 1 investigators. Afatinib versus methotrexate as second-line treatment in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 1): an open-label, randomised phase 3 trial. Lancet Oncol. 2015 May;16(5):583-94. doi: 10.1016/S1470-2045(15)70124-5. Epub 2015 Apr 16. PMID 25892145